CLINICAL TRIAL: NCT04448600
Title: Baha Bone Conduction Implants and Magnetic Resonance Imaging
Brief Title: Bone Conduction Implant and MRI
Acronym: BAHA-IRM
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2019-A03233-54
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Bone Anchored Devices; Osseo-Integrated Implants; MRI Scans; Artifacts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — The patients included in the study will all have a cerebral MRI as part of the cholesteatoma follow-up or for the assessment of cerebral or inner ear pathology.
  - ENT evaluation

SUMMARY:
Bone conduction implants (BCI) are widely used in cases of conductive/ mixed hearing loss or single side deafness when surgical treatment or air hearing aids are not feasible. There are two types of BCI, abutments (which pass through the skin) and magnets (where a subcutaneous magnet is coupled to an external magnet). Pathologies (such as cholesteatoma) leading to the insertion of this hearing implant often require prolonged MRI follow-up. However, both the abutment and the magnet are responsible for imaging artifacts that limit its interpretation. Frequency and extent of these artifacts remain unclear in the literature. In our experience, the magnet, due to its size and composition, produces larger artifacts than the abutment. The main objective of our study is to compare MRI artifacts for each of these device types (abutment and magnet).

DETAILED DESCRIPTION:
The patients included in the study will all have a cerebral MRI as part of the cholesteatoma follow-up or for the assessment of cerebral or inner ear pathology.

* ENT evaluation: The position of the implant will be evaluated. The distance from the external ear canal (center of the abutment or center of the magnet) will be measured on the patient using a ribbon meter. The angle between the implant and the orbital plane (in degrees) will be evaluated on a profile photograph.
* Imaging evaluation: MRI examinations will be anonymized and sent to a single core laboratory for reading. One reader, a board-certified neuroradiologist with 5 years of experience in inner ear imaging, blinded to all data, will review all MRI examinations on a dedicated workstation with the Carestream Vue PACS software (Carestream Health, Rochester, NY). The main outcome measures will be the size of artifacts and the interpretability of sequences. The following MRI sequences will be performed on a 1.5T scanner (1.5T Philips®, Ingenia), covering the temporal bones :

ROUTINE SEQUENCES

* 2D Diffusion weighted-imaging (WI)
* High-resolution 3D T2-WI TSE (DRIVE)
* Post-contrast 2D T1-WI TSE (axial and coronal planes)

ADDITIONAL SEQUENCES (approximately 20 minutes of additional acquisition time) :

* 2D DWI (axial and coronal) phase inverted
* 2D T2-WI TSE (axial and coronal planes)
* High-resolution 3D T2-WI gradient echo (bFFE)
* post contrast 3D T1-WI TSE and gradient echo (THRIVE)

ELIGIBILITY:
Inclusion Criteria Patient over 18 years old Patient with a Baha bone conduction hearing implant, who must perform an MRI examination of the brain, internal auditory canal or middle ear, with or without injection Affiliate or beneficiary of a social security scheme Express consent to participate in the study Exclusion Criteria Patient benefiting from a legal protection measure Pregnant or lactating woman MRI examination not feasible Contraindications to the practice of an MRI: ocular metallic foreign body,certain implanted materials, pacemakers, claustrophobia Contraindications to gadolinium injection, if an MRI is prescribed with gadolinium contrast agent injection allergy, known renal failure: glomerular filtration rate inferior to 30mL by min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a Baha magnet or abutment hearing implant and having to perform a brain MRI.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Artifact size, measured in millimeters, on MRI sequences. | baseline
  mm

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild (FOR), Paris, France

IPD SHARING:
Plan to Share IPD: No